CLINICAL TRIAL: NCT03992521
Title: Breast Cancer Liquid Biopsy Stratification
Acronym: BALIBISTRA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: BreastctDNA01
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Plasma DNA and DNA from primary tumors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Nucleosome positioning — Stratification of patients based on nucleosome positioning from plasma DNA.

SUMMARY:
Breast cancer is the most common cancer in Austrian women. Estimation of prognosis and treatment strategies is increasingly being dependent on stratification of tumors into different entities or classes. Currently, clinical routine stratification of tumors is mostly based on hormone receptor, HER2 status, and estimation of proliferation. However, a more robust and objective classification of tumors can be achieved by elucidation of further biological properties, which is also of increasing significance, as novel anticancer therapies are based on biological mechanisms. Consequently, available information from molecular analyses is increasingly being implemented in routine diagnostic assays with the aim to improve stratification for optimal treatment selection. To date the most extensive molecular-based taxonomy of breast cancer has been achieved by a classification based on combining gene expression and somatic copy number alterations (SCNAs), referred to as integrative clusters. Tissue biopsies are the current gold standard to attain such a classification. However, they can often be difficult to obtain in the metastatic setting and are subject to sampling bias due to intratumor heterogeneity. "Liquid biopsies" are, among other analytes, based on the analysis of cell-free DNA (cfDNA) which contains circulating tumor DNA (ctDNA), i.e. DNA fragments shed from normal and tumor cells into the blood, in patients with cancer. cfDNA can be obtained minimally invasive with a blood draw, allows for the "real time" analysis of tumor DNA from the circulation, and blood samples can be repeated at any time point, which is especially important for monitoring response to therapy. The investigator's group has extensive expertise in the analysis of cfDNA and has developed a plethora of approaches for ctDNA analysis. Recently, the investigators have developed a new approach, which relates to nucleosome positions and gene expression. cfDNA fragments have been associated with the release of DNA from apoptotic cells after enzymatic processing and hence consist mainly of mono-nucleosomal DNA. By performing whole-genome sequencing of cfDNA the investigators could demonstrate that at transcriptional start sites, the nucleosome occupancy results in different read-depth coverage patterns in expressed and silent genes. By employing machine learning for gene classification, the investigators were able to classify genes in cells releasing their DNA into the circulation as expressed. The main hypothesis of the project is that integrative breast cancer clusters can be established from directly blood without the need for an invasive tissue biopsy. Hence, the study aims include refining stratification of patients for an improved selection of treatment strategies. Furthermore, the investigators will obtain novel insights into the biology of metastatic breast cancer, so that this project will have important implications for patients, clinical oncologists, pathologists, pharmacologists, and all basic researchers interested in cancer.

DETAILED DESCRIPTION:
The investigators collected 340 plasma samples from 144 clinically annotated patients with detailed clinical data. All plasma samples were already analyzed by plasma-Seq, an approach, which measures copy number from sequence read depth, for a first evaluation of somatic copy number alterations (SCNAs). As this project represents a feasibility study, the investigators want to evaluate to what extend cis-acting alterations can be determined, i.e. establish the corresponding gene expression changes via nucleosome position mapping as previously published by our group. The results will be corroborated by analyses of the corresponding primary tumor by SCNA-seq and RNA-seq.

From the 340 plasma samples the investigators selected 59 as representative for being either luminal (i.e. those with amplifications at 17q23, 11q13/q14, 8p12, 8q, and gains of 16p and 1q; n=25), basal (i.e. gains of 8q, 10p, 12p and various amplifications occurring due to the high-genomic instability; n=25), and ERBB2/HER2 (i.e. high-level amplification on 17q, centered and including the HER2 gene; n=9). These samples will be sequenced with high coverage (70x) so that both mutations and nucleosome positions can be extracted from the obtained sequences.

ELIGIBILITY:
Inclusion Criteria:

Histological diagnosis of breast cancer, availability of primary tumor tissue and plasma DNA with a high ctDNA content.

Exclusion Criteria:

Patient rejects the participation.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females with breast cancer
Study Population: The study includes women with proven histological diagnosis of breast cancer and appropriate clinical data.
  Participants were recruited at the Medical University Hospital of Graz.
Sampling Method: Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Evaluating as proof-of-concept the ability to stratify patients solely based on a detailed plasma DNA analysis | Three years
  Clinico-pathological characteristics including prior and subsequent therapies were recorded for each patient. For each patient a standard classification into luminal, basal, ERBB2/HER2 was conducted and is available.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Speicher, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ulz P, Thallinger GG, Auer M, Graf R, Kashofer K, Jahn SW, Abete L, Pristauz G, Petru E, Geigl JB, Heitzer E, Speicher MR. Inferring expressed genes by whole-genome sequencing of plasma DNA. Nat Genet. 2016 Oct;48(10):1273-8. doi: 10.1038/ng.3648. Epub 2016 Aug 29. PMID 27571261
- [Background] Heitzer E, Haque IS, Roberts CES, Speicher MR. Current and future perspectives of liquid biopsies in genomics-driven oncology. Nat Rev Genet. 2019 Feb;20(2):71-88. doi: 10.1038/s41576-018-0071-5. PMID 30410101
- [Background] Ulz P, Belic J, Graf R, Auer M, Lafer I, Fischereder K, Webersinke G, Pummer K, Augustin H, Pichler M, Hoefler G, Bauernhofer T, Geigl JB, Heitzer E, Speicher MR. Whole-genome plasma sequencing reveals focal amplifications as a driving force in metastatic prostate cancer. Nat Commun. 2016 Jun 22;7:12008. doi: 10.1038/ncomms12008. PMID 27328849
- [Background] Ulz P, Heitzer E, Speicher MR. Co-occurrence of MYC amplification and TP53 mutations in human cancer. Nat Genet. 2016 Feb;48(2):104-6. doi: 10.1038/ng.3468. No abstract available. PMID 26813759